CLINICAL TRIAL: NCT05649371
Title: A Multiphasic Prehabilitation Exercise Program For Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Multiphasic Prehab Allo-HSCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ACE-HSCT
Record Dates: First submitted 2022-11-07; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-10

CONDITIONS: Leukemia
Keywords: Prehabilitation; Exercise; Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Leukemia; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Hybrid implementation-effectiveness study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental)
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — A multiphasic exercise prehabilitation program for alloHSCT candidates across each treatment phase, that includes behaviour change support

SUMMARY:
The purpose of this study is to implement a prehabilitation intervention to enhance recovery for people undergoing allogeneic stem cell transplant for hematologic malignancies. All participants in this study will receive a prehabilation intervention in addition to usual care (no change to their chemotherapy protocols or transplant) and several quality of life and fitness scores will be measured throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years or older, undergoing an allo-HSCT for acute leukemia.
* Approval to engage in exercise as per screening by the CSEP or ACSM certified CEP and/or clinician
* Ability to provide written informed consent and understand study information.

Exclusion Criteria:

* Less than 18 years old
* Diagnosed with acute leukemia but not undergoing work-up for allo-HSCT
* Unable to read/communicate in English (i.e., unable to complete experimental procedures such as patient-reported outcomes).
* Neurological or musculoskeletal comorbidity inhibiting exercise.
* Diagnosed psychotic, addictive, or major cognitive disorders.
* Severe coronary artery disease (Canadian Cardiovascular Society class III or greater).
* Significant congestive heart failure (New York Heart Association class III or greater).
* Severe thrombocytopenia (platelets <10) - ok if transfused platelets prior to exercise.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementing an Exercise Program for Patients Undergoing Allogeneic-HSCT, Measured by Participant Attendance | 6-9 months
  Review participant attendance/participation in the program and the questionnaires.

SECONDARY OUTCOMES:
Amount of Physical Activity Measured With Activity Tracker | 6-9 months
  Quantity of physical activity, measured in hours.
Exercise Behaviour Measured with Modified Godin Leisure Time Exercise Questionnaire | 6-9 months
  Self reported measure of physical activity. Higher scores are better.
Patient Quality of Life Measured with the Functional Assessment of Cancer Therapy-Bone Marrow Transplant and EuroQol 5 Dimension 5 Level Questionnaire | 6-9 months
  Self reported physical, emotional and functional well-being.
Level of Fatigue Measured with the Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) Questionnaire | 6-9 months
  Self reported level of fatigue during daily activities. Lower scores mean less fatigue.
Amount of Anxiety and depression Measured with the Hospital Anxiety and Depression Scale (HADS) Questionnaire | 6-9 months
  Self reported level of anxiety and depression. Higher scores indicate more anxiety and depression.
Amount of Symptom burden Measured with the Edmonton Symptom Assessment System-revised (ESAS-r) Questionnaire | 6-9 months
  Self reported symptoms. Higher scores indicate more symptoms.
Patient's Performance Status Measured by the Eastern Cooperative Oncology Group (ECOG) Scale | 6-9 months
  Objective score of patient's level of functioning. Lower scores indicate better functioning.
Handgrip Strength Measured by Handgrip Dynamometry | 6-9 months
  Maximum isometric strength of the hand and forearm muscles.
Balance Measured by Single Leg Stance Test | 6-9 months
  Static postural and balance control, measured in seconds.
Lower Limb Muscular Endurance Measured with 30-second sit-to-stand Test | 6-9 months
  Tests leg strength and endurance, measured in number of stands in 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Culos-Reed, PhD, Study Director — Health and Wellness Lab and the Thrive Centre